CLINICAL TRIAL: NCT01136343
Title: Comparison of Predictive Factors Related to Coronary Artery Disease Among Different Menopausal Status and Effect of a Life Style Management Program on Risk Factors Modification Among Middle-aged Women
Brief Title: Comparison of Predictive Factors Related to Coronary Artery Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Medical University WanFang Hospital (Other)
Responsible Party: Principal Investigator, Chii Jeng, Taipei Medical University, Taipei Medical University WanFang Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 99001
Record Dates: First submitted 2010-05-31; First posted 2010-06-03 (Estimated); Last update posted 2023-03-22 (Actual); Status verified 2023-03

CONDITIONS: Coronary Artery Disease
Keywords: women; middle age; risk factor
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- lifestyle modified project (Experimental): education, counseling
  Interventions: Other: lifestyle modified project
- control (No Intervention): waiting list control

INTERVENTIONS:
Other: lifestyle modified project — education, counseling
  Arms: lifestyle modified project

SUMMARY:
In Taiwan, heart disease and cerebrovascular disease ranked the second and third of ten leading causes of death in female in 2007; half of these deaths is due to coronary artery disease (CAD). Postmenopausal status is an independent risk factor for CAD. Early assessment and proper management of risk factors may reduce the prevalence rate of CAD. In the past decade, despite increased attention to CAD in women, most studies focused on certain menopausal status instead of all phases of menopause or on risk factors limited to related metabolic syndrome. Because the prevalence of risk factors related to CAD is influenced by various physiological and lifestyle status in different menopausal statuses, the purpose of this study, at the first stage, is to explore respectively the risk factors of CAD among middle-aged women in three menopausal statuses. At the second stage, the influence of a lifestyle management program on risk factors modification among pre-menopausal women is examined in this study.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of CAD by coroangiography
* LVEF >30%

Exclusion Criteria:

* impairment of physical activity
* history of psychiatric disorder, vital arrhythmia

Ages: 40 Years to 64 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 130 (Actual)
Dates: Start 2010-02; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
lifestyle
  physical activity, dietary, depression, anxiety

SECONDARY OUTCOMES:
metabolic | 6 months
  blood pressure, lipid profile, blood sugar, obesity
biomarkers
  hsCRP, homocysteine, leptin

CONTACTS AND LOCATIONS:
Overall Officials: Chii Jeng, Principal Investigator — Taipei Medical University College of Nursing
Locations (1):
- Wan Fang Hospital, Taipei, Taiwan